CLINICAL TRIAL: NCT03162614
Title: Efficacy, Immunogenicity and Safety Study of GSK Biologicals' Candidate Malaria Vaccine (SB257049) Evaluating Various Dose Schedules in a Sporozoite Challenge Model in Healthy Malaria-naïve Adults
Brief Title: Efficacy, Immunogenicity and Safety Study of GSK Biologicals' Candidate Malaria Vaccine Evaluating Different Dose Schedules in a Sporozoite Challenge Model in Healthy Malaria-naïve Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205081
Record Dates: First submitted 2017-05-15; First posted 2017-05-22 (Actual); Results first posted 2019-07-24 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Malaria
Keywords: healthy volunteers; Malaria; malaria vaccine; controlled human challenge; RTS,S/AS01
MeSH Terms: conditions — Malaria | interventions — RTS malaria vaccine; RTS,S-AS01B vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- AduFx Group (Active Comparator): Healthy subjects, between, and including, 18 and 55 years of age, who received RTS,S/AS01B full dose at Month 0 and Month 1 and 1/5th of RTS,S/AS01B full dose at Month 7, and underwent sporozoite challenge.
  Interventions: Biological: RTS,S/AS01B; Procedure: Sporozoite-infected mosquitoes challenge.
- 2PedFx Group (Experimental): Healthy subjects, between, and including, 18 and 55 years of age, who received RTS,S/AS01E double dose at Month 0 and Month 1, and 1/5th of double dose RTS,S/AS01E at Month 7, and underwent sporozoite challenge.
  Interventions: Biological: RTS,S/AS01E; Procedure: Sporozoite-infected mosquitoes challenge.
- PedFx Group (Experimental): Healthy subjects, between, and including, 18 and 55 years of age, who received RTS,S/AS01E full dose at Month 0 and Month 1, and 1/5th of RTS,S/AS01E full dose at Month 7, and underwent sporozoite challenge.
  Interventions: Biological: RTS,S/AS01E; Procedure: Sporozoite-infected mosquitoes challenge.
- Adu2Fx Group (Experimental): Healthy subjects, between, and including, 18 and 55 years of age, who received RTS,S/AS01B full dose at Month 0 and 1/5th of RTS,S/AS01B full dose at Month 1 and Month 7, and underwent sporozoite challenge.
  Interventions: Biological: RTS,S/AS01B; Procedure: Sporozoite-infected mosquitoes challenge.
- Adu1Fx Group (Active Comparator): Healthy subjects, between, and including, 18 and 55 years of age, who received RTS,S/AS01B full dose at Month 0 and 1/5th of RTS,S/AS01B full dose administered at Month 7, and underwent sporozoite challenge.
  Interventions: Biological: RTS,S/AS01B; Procedure: Sporozoite-infected mosquitoes challenge.
- Control Group (Other): Healthy subjects, between, and including, 18 and 55 years of age, who did not receive any immunization but underwent sporozoite challenge.
  Interventions: Procedure: Sporozoite-infected mosquitoes challenge.

INTERVENTIONS:
Biological: RTS,S/AS01E — Subjects will receive intramuscular injection of RTS,S/AS01E.
  Arms: 2PedFx Group; PedFx Group
Biological: RTS,S/AS01B — Subjects will receive intramuscular injection of RTS,S/AS01B.
  Arms: Adu1Fx Group; Adu2Fx Group; AduFx Group
Procedure: Sporozoite-infected mosquitoes challenge. — Mosquitoes infected approximately 2-3 weeks earlier that are likely to contain sporozoites in their salivary glands will be allowed to feed on the subjects. For each subject, five mosquitoes will be allowed to feed over five minutes, after which they will be dissected to confirm how many were infected, and the salivary glands scored. If required additional mosquitoes will be allowed to feed until a total of five infected mosquitoes with a minimum of 2+ salivary gland scores have fed.
  The challenge occurs approximately 90 days (three months) after the last vaccination.
  Subjects will be monitored during 28 days after having bitten by mosquitoes and when parasites are found in their blood, they will be treated with appropriate anti-malarial drugs.

SUMMARY:
This study is designed to evaluate efficacy, immunogenicity and safety of various dose schedules of GSK Biologicals' candidate malaria vaccines RTS,S/AS01B (adult formulation) and RTS,S/AS01E (pediatric formulation) in healthy malaria-naïve subjects aged 18-55 years. The purpose of this study is to investigate whether changes in dosing schedule are associated with increased or equivalent protection, and to evaluate the immune mechanisms associated with vaccine efficacy under varying dosing schedules.

DETAILED DESCRIPTION:
Protocol Amendment 1 incorporated: additional blood sampling for assessment of parasitemia (polymerase chain reaction [PCR] testing); clarification that blood samples for both peripheral blood mononuclear cells (PBMC) and plasma will be collected for repository storage; revision of volume of whole blood samples to be taken for parasitemia assessment; clarification that urine pregnancy tests will be conducted for all females and not just those of childbearing potential; deletion of visit at Day 1 post day of challenge; clarification that RNA sequencing and not deep sequencing will be performed in this study.

Note that as a result of internal change in data standards terminology, the study data collected was converted to cDISC and the statistical analysis plan was amended accordingly. "Day 0" in the study design was replaced by "Day 1"; consequently, "Day n" was replaced by "Day n+1". Thus, the timeframes (Day 0, Day n) of Outcome Measures described in this study record are different to that denoted in the full protocol document posted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing of any study specific procedure.
* A male or female between, and including, 18 and 55 years of age at the time of enrolment.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Available to participate for the duration of the study.
* Female subjects of non-childbearing potential may be enrolled in the study.

  - Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test at enrolment, and
  * has agreed to continue adequate contraception during the entire treatment period and for two months after completion of the vaccination series and/or malaria challenge.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines during the period starting 30 days before the first dose of study vaccines (Day -29 to Day 0), or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Chronic use of antibiotics with antimalarial effects.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting seven days before the first dose.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Documented HIV-positive subject.
* Previous vaccination against malaria.
* History of malaria chemoprophylaxis within 60 days prior to vaccination.
* Any history of malaria (for the vaccine groups).
* Planned travel to malaria endemic areas during the study period.
* History of splenectomy.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* History of anaphylaxis post-vaccination.
* Hypersensitivity to latex.
* History of any reaction or hypersensitivity likely to be exacerbated by chloroquine.
* History of psoriasis and porphyria, which may be exacerbated after chloroquine treatment.
* Current use of medications known to cause drug reactions to chloroquine.
* History of severe reactions to mosquito bites.
* Major congenital defects.
* Serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment. Fever is defined as temperature ≥ 37.5°C/99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C/100.4°F for rectal route.

  - Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Any abnormal baseline laboratory screening tests: alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine, hemoglobin, platelet count, total white blood cells (WBC), out of normal range as defined in the protocol.
* Evidence of increased cardiovascular disease risk, "moderate" or "high", according to the National health and nutrition examination survey I criteria.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Personal history of autoimmune disease.
* Administration of immunoglobulins and/or any blood products during the period starting three months before the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of blood donation within 56 days preceding enrolment.
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20719

REFERENCES:
- [Background] James E. Moon, Christian Ockenhouse, Jason A. Regules, Johan Vekemans, Cynthia Lee, Ilin Chuang, Magali Traskine, Erik Jongert, Karen Ivinson, Danielle Morelle, Jack L. Komisar, Marc Lievens, Martha Sedegah, Lindsey Garver, April K. Sikaffy, Norman C. Waters, William Ripley Ballou, Opokua Ofori-Anyinam for the RTS,S Malaria Vaccine Working Group. CLI_092_A Phase IIa Controlled Human Malaria Infection and Immunogenicity Study of RTS,S/AS01E and RTS,S/AS01B Delayed Fractional Dose Regimens in Malaria-Naïve Adults. J Infect Dis. 2020 Jul 20;jiaa421. doi: 10.1093/infdis/jiaa421. Online ahead of print.
- [Derived] Spreng RL, Seaton KE, Lin L, Hilliard S, Horn GQ, Abraha M, Deal AW, Li K, Carnacchi AJ, Feeney E, Shabbir S, Zhang L, Bekker V, Mudrak SV, Dutta S, Mercer LD, Gregory S, King CR, Wille-Reece U, Jongert E, Kisalu NK, Tomaras GD, Dennison SM. Identification of RTS,S/AS01 vaccine-induced humoral biomarkers predictive of protection against controlled human malaria infection. JCI Insight. 2024 Oct 8;9(19):e178801. doi: 10.1172/jci.insight.178801. PMID 39377226
- [Derived] Moon JE, Ockenhouse C, Regules JA, Vekemans J, Lee C, Chuang I, Traskine M, Jongert E, Ivinson K, Morelle D, Komisar JL, Lievens M, Sedegah M, Garver LS, Sikaffy AK, Waters NC, Ballou WR, Ofori-Anyinam O; RTS,S Malaria Vaccine Working Group. A Phase IIa Controlled Human Malaria Infection and Immunogenicity Study of RTS,S/AS01E and RTS,S/AS01B Delayed Fractional Dose Regimens in Malaria-Naive Adults. J Infect Dis. 2020 Oct 13;222(10):1681-1691. doi: 10.1093/infdis/jiaa421. PMID 32687161

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
Started | 26 | 26 | 26 | 26 | 26 | 24
Completed | 20 | 21 | 22 | 19 | 21 | 24
Not Completed | 6 | 5 | 4 | 7 | 5 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1 | 0 | 0
Not completed — Missed vaccination, exclusion criteria | 2 | 2 | 2 | 4 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group | Total
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 24 | 154
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (8.4) | 30.8 (9.6) | 32.0 (10.4) | 32.4 (10.9) | 32.2 (10.3) | 34.6 (11.9) | 32.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 12 | 4 | 10 | 10 | 57
  Male | 15 | 16 | 14 | 22 | 16 | 14 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 3 | 2 | 2 | 1 | 0 | 9
  Black Or African American | 8 | 6 | 10 | 9 | 7 | 8 | 48
  Native Hawaiian Or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Other, Not Specified | 0 | 1 | 2 | 2 | 4 | 1 | 10
  White | 17 | 16 | 12 | 13 | 14 | 14 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Occurrence of Plasmodium Falciparum (P. Falciparum) Parasitemia for Each Vaccination Schedule Versus Infectivity Controls
Description: Occurrence of P. falciparum parasitemia (defined by a positive blood slide) following sporozoite challenge. Post-challenge, parasitemia was determined by microscopy of Giemsa-stained thick blood films (smear). Microscopy was performed on thick smears using a validated standard operation procedure. For the analysis of proportion affected (relative risk), all subjects included in the analysis were considered at risk of infection and no censoring or elimination was applied for subjects not completing the entire protocol defined post challenge follow-up (Day 315 - 28 days post challenge).
Time Frame: Following sporozoite challenge starting 3 months after the last vaccine dose (Day 287) for up to 28 days post-challenge (Day 315).
Population: Analysis was performed on Per-Protocol Set, which included all subjects fulfilling eligibility criteria who received vaccinations according to protocol procedures, did not report any underlying medical condition influencing the efficacy response, had available data concerning immunogenicity outcome measures, and underwent P. falciparum challenge.
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
Number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 22
Participants | 9 | 5 | 8 | 9 | 15 | 22
Statistical Analysis 1: Comparison: AduFx Group vs Control Group; Efficacy analysis aimed at comparing RTS,S/AS01B administered as full doses at Month 0 and Month 1 and 1/5th dose at Month 7 (AduFx Group versus Control Group); Test type: Other — Vaccine efficacy rate was calculated as 100*(1-RR) with RR=relative risk of developing the disease for vaccinated people compared to unvaccinated people; p < .001, Fisher Exact; Vaccine efficacy rate = 55, 95% CI 2-sided [27 to 72]
Statistical Analysis 2: Comparison: 2PedFx Group vs Control Group; Efficacy analysis aimed at comparing RTS,S/AS01E administered as double full doses at Month 0 and Month 1 and 1/5th double dose at Month 7 (2Ped Fx Group versus Control Group); Test type: Other — [test comment as in outcome 1, analysis 1]; p < .001, Fisher Exact; Vaccine efficacy rate = 76, 95% CI 2-sided [49 to 89]
Statistical Analysis 3: Comparison: PedFx Group vs Control Group; Efficacy analysis aimed at comparing RTS,S/AS01E administered as full doses at Month 0 and Month 1 and 1/5th dose at Month 7 (PedFx Group versus Control Group); Test type: Other — [test comment as in outcome 1, analysis 1]; p < .001, Fisher Exact; Vaccine efficacy rate = 64, 95% CI 2-sided [37 to 79]
Statistical Analysis 4: Comparison: Adu2Fx Group vs Control Group; Efficacy analysis aimed at comparing RTS,S/AS01B administered as full dose at Month 0 and 1/5th dose at Month 1 and Month 7 (Adu2Fx Group versus Control Group); Test type: Other — [test comment as in outcome 1, analysis 1]; p < .001, Fisher Exact; Vaccine efficacy rate = 55, 95% CI 2-sided [27 to 72]
Statistical Analysis 5: Comparison: Adu1Fx Group vs Control Group; Efficacy analysis aimed at comparing RTS,S/AS01B administered as full dose at Month 0 and 1/5th dose at Month 7 (Adu1Fx Group versus Control Group); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.009, Fisher Exact; Vaccine efficacy rate = 29, 95% CI 2-sided [6 to 46]

2. Secondary Outcome: Time to Onset of P. Falciparum Parasitemia After Sporozoite Challenge for Each Vaccination Schedule
Description: For the analyses of time to onset of parasitemia, time at risk started on first day of challenge. Time at risk was censored on Day 315 (28 days post challenge), drop-out date, start date of antimalarial treatment or date meeting an endpoint, whichever occurs first.
Time Frame: Following sporozoite challenge starting 3 months after the last vaccine dose (at Day 287) for up to 28 days post-challenge (at Day 315).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
Number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 22
Days | 14.8 (1.2) | 14.6 (1.1) | 14.3 (2.0) | 14.9 (2.1) | 14.2 (2.4) | 12.7 (1.9)

3. Secondary Outcome: Anti-Circumsporozoite (Anti-CS) Repeat Region Antibody Concentrations
Description: Anti-CS antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in Enzyme-linked immunosorbent assay Unit per milliliter (EU/mL). The cut-off for the assay was 1.9 EU/mL. The GMC calculations were performed by taking the anti-log of the mean of the log transformations (base 10). Antibody concentrations below the cut-off of the assay were given an arbitrary value of half the cut-off (=1.0) for the purpose of GMC calculation.
Time Frame: At Day 1, Day 59, Day 197, Day 227, Day 287, Day 315, and Day 377 for subjects from AduFx, 2PedFx, PedFx, and Adu2Fx Groups. At Day 1, Day 197, Day 227, Day 287, Day 315, and Day 377 for subjects from Adu1Fx Group
Population: Analysis was performed on subjects fulfilling eligibility criteria, who received study vaccination according to protocol procedures (therefore, not on subjects from the Control Group), did not report any medical condition influencing the efficacy response, had data concerning immunogenicity outcome measures, and underwent P. falciparum challenge.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group
Number analyzed (Participants) | 20 | 21 | 22 | 20 | 21
EU/mL
  At Day 1 | 1 [1.0 to 1.0] | 1 [1.0 to 1.0] | 1 [1.0 to 1.0] | 1 [1.0 to 1.0] | 1 [1.0 to 1.0]
  At Day 59: number analyzed (Participants) | 20 | 21 | 22 | 20 | 0
  At Day 59 | 108.2 [70.1 to 167.0] | 107.8 [73.0 to 159.1] | 53.8 [39.0 to 74.1] | 61.7 [47.6 to 79.9] |
  At Day 197 | 30 [17.9 to 50.5] | 39.3 [23.8 to 64.8] | 15.1 [9.3 to 24.5] | 19.4 [13.2 to 28.5] | 3.8 [2.0 to 7.2]
  At Day 227 | 85.9 [50.8 to 145.5] | 79.8 [54.7 to 116.6] | 50.2 [35.5 to 70.9] | 64 [42.8 to 95.8] | 22.1 [12.0 to 40.8]
  At Day 287 | 61.4 [34.7 to 108.8] | 57.6 [38.2 to 87.1] | 34.4 [23.1 to 51.1] | 38.1 [20.8 to 69.9] | 12.3 [6.2 to 24.4]
  At Day 315 | 56.6 [32.5 to 98.4] | 51 [33.3 to 78.0] | 31.3 [21.2 to 46.3] | 44.1 [27.8 to 70.1] | 10.6 [5.2 to 21.5]
  At Day 377: number analyzed (Participants) | 20 | 20 | 22 | 19 | 20
  At Day 377 | 43.7 [24.9 to 76.8] | 38.1 [24.3 to 59.8] | 25 [16.5 to 37.9] | 31.7 [19.6 to 51.3] | 9.5 [4.8 to 19.0]

4. Secondary Outcome: Anti-Hepatitis B (Anti-HBs) Immunoglobulin G (IgG) Antibody Concentrations
Description: Anti-HBs IgG antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in milli-International Unit per milliliter (mIU/ml). The cut-off for the assay was 6.2 mIU/mL.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group
Number analyzed (Participants) | 20 | 21 | 22 | 20 | 21
mIU/mL
  At Day 1: number analyzed (Participants) | 20 | 21 | 21 | 20 | 21
  At Day 1 | 44.1 [15.6 to 124.3] | 68.8 [20.4 to 231.7] | 45.7 [15.2 to 137.5] | 21.8 [9.0 to 52.6] | 16 [6.5 to 39.6]
  At Day 59: number analyzed (Participants) | 20 | 21 | 20 | 20 | 0
  At Day 59 | 42616.7 [12325.1 to 147356.7] | 28894.8 [8705.8 to 95903.3] | 26149.3 [8588.7 to 79615.2] | 14710.6 [3837.0 to 56398.8] |
  At Day 197: number analyzed (Participants) | 20 | 21 | 21 | 20 | 21
  At Day 197 | 19369.3 [8325.5 to 45062.6] | 15358.8 [5971.2 to 39505.1] | 11269.1 [4892.1 to 25958.8] | 6846.7 [2273.5 to 20618.8] | 2031.7 [715.9 to 5766.4]
  At Day 227 | 45959.9 [27093.8 to 77962.8] | 30994.5 [15352.8 to 62572.4] | 28560.6 [15532.4 to 52516.4] | 26717 [12916.3 to 55263.3] | 35620.9 [22337.4 to 56803.7]
  At Day 287: number analyzed (Participants) | 20 | 21 | 22 | 19 | 21
  At Day 287 | 36266.3 [21828.7 to 60252.9] | 20712.2 [10050.4 to 42684.5] | 19126.1 [9889.0 to 36991.5] | 13911.3 [4939.4 to 39179.9] | 16376.8 [9798.1 to 27372.8]
  At Day 315: number analyzed (Participants) | 20 | 21 | 22 | 19 | 21
  At Day 315 | 33027.7 [19159.7 to 56933.4] | 18527.8 [8862.8 to 38732.5] | 17465.5 [8798.2 to 34671.2] | 16685 [8192.0 to 33982.9] | 12609.9 [7499.3 to 21203.5]
  At Day 377: number analyzed (Participants) | 20 | 20 | 21 | 19 | 20
  At Day 377 | 27823 [15910.1 to 48655.8] | 15083.7 [6953.8 to 32718.4] | 13716 [6456.7 to 29136.9] | 11257.6 [5164.7 to 24538.5] | 10975.2 [5889.9 to 20451.3]

5. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Solicited local symptoms assessed are pain, redness and swelling. Any occurrence of symptom regardless of intensity grade. Any Redness or any Swelling symptom = any symptom greater than (>) 0 millimeter (mm).
Time Frame: Within the 7-day period (Days 1-7) after dose 1, dose 2 (except for Adu1Fx Group) and dose 3.
Population: The analysis was performed on Intent-To-Treat Set, which included all subjects who received at least one dose of study vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 25
Participants
  Pain, dose 1 | 23 | 21 | 22 | 22 | 19
  Redness, dose 1 | 8 | 11 | 4 | 8 | 9
  Swelling, dose 1 | 5 | 12 | 3 | 4 | 5
  Pain, dose 2: number analyzed (Participants) | 26 | 25 | 26 | 26 | 0
  Pain, dose 2 | 20 | 16 | 20 | 12 |
  Redness, dose 2: number analyzed (Participants) | 26 | 25 | 26 | 26 | 0
  Redness, dose 2 | 8 | 10 | 5 | 4 |
  Swelling, dose 2: number analyzed (Participants) | 26 | 25 | 26 | 26 | 0
  Swelling, dose 2 | 5 | 8 | 6 | 3 |
  Pain, dose 3: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23
  Pain, dose 3 | 11 | 12 | 13 | 16 | 15
  Redness, dose 3: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23
  Redness, dose 3 | 7 | 10 | 10 | 11 | 6
  Swelling, dose 3: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23
  Swelling, dose 3 | 3 | 6 | 5 | 3 | 3

6. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Solicited general symptoms assessed are fatigue, gastrointestinal symptoms, headache and fever. Any occurrence of symptom regardless of intensity grade. Fever was defined as temperature equal or greater than (≥) 37.5 degrees Celsius (°C) for oral route, axillary or tympanic route or 38.0°C for rectal route.
Time Frame: Within the 7-day period (Days 1-7) after dose 1, dose 2 (except for Adu1Fx Group) and dose 3.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 25
Participants
  Fatigue, dose 1 | 13 | 14 | 13 | 10 | 11
  Gastrointestinal symptoms, dose 1 | 5 | 8 | 5 | 4 | 6
  Headache, dose 1 | 15 | 14 | 10 | 12 | 9
  Fever, dose 1 | 3 | 6 | 2 | 3 | 3
  Fatigue, dose 2: number analyzed (Participants) | 26 | 25 | 26 | 26 | 0
  Fatigue, dose 2 | 11 | 12 | 10 | 6 |
  Gastrointestinal symptoms, dose 2: number analyzed (Participants) | 26 | 25 | 26 | 26 | 0
  Gastrointestinal symptoms, dose 2 | 3 | 6 | 7 | 3 |
  Headache, dose 2: number analyzed (Participants) | 26 | 25 | 26 | 26 | 0
  Headache, dose 2 | 13 | 14 | 11 | 6 |
  Fever, dose 2: number analyzed (Participants) | 26 | 25 | 26 | 26 | 0
  Fever, dose 2 | 6 | 6 | 3 | 1 |
  Fatigue, dose 3: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23
  Fatigue, dose 3 | 4 | 6 | 8 | 11 | 8
  Gastrointestinal symptoms, dose 3: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23
  Gastrointestinal symptoms, dose 3 | 4 | 2 | 6 | 0 | 5
  Headache, dose 3: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23
  Headache, dose 3 | 6 | 7 | 6 | 9 | 9
  Fever, dose 3: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23
  Fever, dose 3 | 0 | 2 | 0 | 2 | 0

7. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) After Any Vaccination
Description: An unsolicited adverse event is any untoward medical occurrence in a clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited adverse event is any event reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 30-day period (Days 1-30), after any vaccination (across doses)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26
Participants | 18 | 18 | 15 | 17 | 10

8. Secondary Outcome: Number of Subjects With Any Unsolicited AEs After Challenge
Description: An adverse event is any untoward medical occurrence in a clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within the 30-day (Days 1-30) period post-challenge
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Subjects With Any, Fatal or Related Serious Adverse Events (SAEs) After Each Vaccination
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Within the 30-day period (Days 1-30) after any vaccination (across doses)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26
Participants | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Subjects With Any, Fatal or Related SAEs During the Whole Study Period
Description: as for outcome 9
Time Frame: From Day 1 up to study conclusion (Day 377)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Subjects With Any AE and SAE Leading to Withdrawal From Further Vaccination
Description: An adverse event is any untoward medical occurrence in a clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. SAEs include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 1 up to study conclusion (Day 377)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Subjects With Potential Immune Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From Day 1 up to study conclusion (Day 377)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Subjects With Meningitis
Description: Meningitis is to be reported as an adverse event of specific interest and tabulated per study group.
Time Frame: From Day 1 up to study conclusion (Day 377)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Subjects With Abnormal Laboratory Values Gradings
Description: Biochemistry (Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST] and creatinine) and hematological (hemoglobin, platelets, White Blood Cells [WBC] decrease and WBC increase) laboratory values were presented according to toxicity grading scales (Grade 0 [GR0], Grade 1 [GR1], Grade 2 [GR2] Grade 3 [GR3]) and tabulated by group. Grading scale is taken from the [FDA guidance for industry: toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (September 2007)].
Time Frame: At Visit 1 Screening (Day -89 to Day 1), Day 36, Day 59, Day 204, Day 227, between Day 292 & Day 313, and Day 315 for each vaccinated subject.For Infectivity Control subjects at Visit 1b Screening (Day 231 to Day 287),between Day 292 & Day 313,and Day 315
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 24
Participants
  Alanine Aminotransferase, SCR, Gr0 | 25 | 24 | 25 | 25 | 26 | 24
  Alanine Aminotransferase, SCR, Gr1 | 1 | 2 | 1 | 0 | 0 | 0
  Alanine Aminotransferase, SCR, Gr2 | 0 | 0 | 0 | 1 | 0 | 0
  Alanine Aminotransferase, D36, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Alanine Aminotransferase, D36, Gr0 | 26 | 24 | 25 | 25 |  |
  Alanine Aminotransferase, D36, Gr1: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Alanine Aminotransferase, D36, Gr1 | 0 | 1 | 0 | 1 |  |
  Alanine Aminotransferase, D59, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Alanine Aminotransferase, D59, Gr0 | 26 | 24 | 24 | 24 |  |
  Alanine Aminotransferase, D59, Gr1: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Alanine Aminotransferase, D59, Gr1 | 0 | 1 | 1 | 2 |  |
  Alanine Aminotransferase, D204, Gr0: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  Alanine Aminotransferase, D204, Gr0 | 21 | 22 | 24 | 24 | 20 |
  Alanine Aminotransferase, D204, Gr1: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  Alanine Aminotransferase, D204, Gr1 | 2 | 2 | 0 | 1 | 3 |
  Alanine Aminotransferase, D227, Gr0: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Alanine Aminotransferase, D227, Gr0 | 22 | 20 | 23 | 23 | 22 |
  Alanine Aminotransferase, D227, Gr1: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Alanine Aminotransferase, D227, Gr1 | 1 | 2 | 1 | 1 | 1 |
  Alanine Aminotransferase, D227, Gr2: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Alanine Aminotransferase, D227, Gr2 | 0 | 1 | 0 | 0 | 0 |
  Alanine Aminotransferase, D292, Gr0: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Alanine Aminotransferase, D292, Gr0 | 9 | 4 | 7 | 8 | 10 | 22
  Alanine Aminotransferase, D292, Gr1: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Alanine Aminotransferase, D292, Gr1 | 0 | 0 | 1 | 1 | 5 | 0
  Alanine Aminotransferase, D292, Gr2: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Alanine Aminotransferase, D292, Gr2 | 0 | 1 | 0 | 0 | 0 | 1
  Alanine Aminotransferase, D315, Gr0: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  Alanine Aminotransferase, D315, Gr0 | 16 | 20 | 18 | 18 | 18 | 21
  Alanine Aminotransferase, D315, Gr1: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  Alanine Aminotransferase, D315, Gr1 | 3 | 1 | 4 | 2 | 2 | 3
  Alanine Aminotransferase, D315, Gr2: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  Alanine Aminotransferase, D315, Gr2 | 1 | 0 | 0 | 0 | 1 | 0
  Aspartate Aminotransferase, SCR, Gr0 | 26 | 25 | 25 | 25 | 26 | 23
  Aspartate Aminotransferase, SCR, Gr1 | 0 | 1 | 1 | 1 | 0 | 1
  Aspartate Aminotransferase, D36, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Aspartate Aminotransferase, D36, Gr0 | 26 | 25 | 24 | 26 |  |
  Aspartate Aminotransferase, D36, Gr1: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Aspartate Aminotransferase, D36, Gr1 | 0 | 0 | 1 | 0 |  |
  Aspartate Aminotransferase, D59, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Aspartate Aminotransferase, D59, Gr0 | 26 | 24 | 24 | 25 |  |
  Aspartate Aminotransferase, D59, Gr1: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Aspartate Aminotransferase, D59, Gr1 | 0 | 1 | 1 | 1 |  |
  Aspartate Aminotransferase, D204, Gr0: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  Aspartate Aminotransferase, D204, Gr0 | 22 | 23 | 24 | 25 | 22 |
  Aspartate Aminotransferase, D204, Gr1: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  Aspartate Aminotransferase, D204, Gr1 | 1 | 1 | 0 | 0 | 1 |
  Aspartate Aminotransferase, D227, Gr0: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Aspartate Aminotransferase, D227, Gr0 | 23 | 22 | 23 | 23 | 22 |
  Aspartate Aminotransferase, D227, Gr1: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Aspartate Aminotransferase, D227, Gr1 | 0 | 0 | 1 | 0 | 1 |
  Aspartate Aminotransferase, D227, Gr2: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Aspartate Aminotransferase, D227, Gr2 | 0 | 1 | 0 | 1 | 0 |
  Aspartate Aminotransferase, D292, Gr0: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Aspartate Aminotransferase, D292, Gr0 | 9 | 4 | 7 | 9 | 13 | 22
  Aspartate Aminotransferase, D292, Gr1: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Aspartate Aminotransferase, D292, Gr1 | 0 | 0 | 1 | 0 | 2 | 0
  Aspartate Aminotransferase, D292, Gr2: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Aspartate Aminotransferase, D292, Gr2 | 0 | 0 | 0 | 0 | 0 | 1
  Aspartate Aminotransferase, D292, Gr3: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Aspartate Aminotransferase, D292, Gr3 | 0 | 1 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, D315, Gr0: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  Aspartate Aminotransferase, D315, Gr0 | 20 | 21 | 21 | 18 | 20 | 24
  Aspartate Aminotransferase, D315, Gr1: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  Aspartate Aminotransferase, D315, Gr1 | 0 | 0 | 1 | 2 | 1 | 0
  Creatinine, SCR, Gr0 | 26 | 26 | 26 | 25 | 26 | 24
  Creatinine, SCR, Gr1 | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine, D36, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Creatinine, D36, Gr0 | 25 | 25 | 25 | 26 |  |
  Creatinine, D36, Gr1: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Creatinine, D36, Gr1 | 1 | 0 | 0 | 0 |  |
  Creatinine, D59, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Creatinine, D59, Gr0 | 26 | 25 | 25 | 26 |  |
  Creatinine, D204, Gr0: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  Creatinine, D204, Gr0 | 23 | 24 | 24 | 25 | 22 |
  Creatinine, D204, Gr1: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  Creatinine, D204, Gr1 | 0 | 0 | 0 | 0 | 1 |
  Creatinine, D227, Gr0: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Creatinine, D227, Gr0 | 23 | 23 | 24 | 24 | 22 |
  Creatinine, D227, Gr1: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Creatinine, D227, Gr1 | 0 | 0 | 0 | 0 | 1 |
  Creatinine, D292, Gr0: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Creatinine, D292, Gr0 | 9 | 5 | 8 | 8 | 15 | 22
  Creatinine, D292, Gr1: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Creatinine, D292, Gr1 | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine, D292, UNK: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Creatinine, D292, UNK | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine, D315, Gr0: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  Creatinine, D315, Gr0 | 20 | 21 | 21 | 20 | 20 | 24
  Creatinine, D315, Gr1: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  Creatinine, D315, Gr1 | 0 | 0 | 1 | 0 | 1 | 0
  Hemoglobin, SCR, Gr0 | 26 | 26 | 26 | 26 | 26 | 23
  Hemoglobin, SCR, Gr1 | 0 | 0 | 0 | 0 | 0 | 1
  Hemoglobin, D36, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Hemoglobin, D36, Gr0 | 23 | 24 | 22 | 25 |  |
  Hemoglobin, D36, Gr1: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Hemoglobin, D36, Gr1 | 3 | 1 | 3 | 1 |  |
  Hemoglobin, D59, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Hemoglobin, D59, Gr0 | 25 | 25 | 24 | 25 |  |
  Hemoglobin, D59, Gr1: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Hemoglobin, D59, Gr1 | 1 | 0 | 1 | 1 |  |
  Hemoglobin, D204, Gr0: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  Hemoglobin, D204, Gr0 | 20 | 24 | 21 | 25 | 23 |
  Hemoglobin, D204, Gr1: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  Hemoglobin, D204, Gr1 | 3 | 0 | 3 | 0 | 0 |
  Hemoglobin, D227, Gr0: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Hemoglobin, D227, Gr0 | 19 | 23 | 23 | 23 | 23 |
  Hemoglobin, D227, Gr1: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Hemoglobin, D227, Gr1 | 4 | 0 | 1 | 1 | 0 |
  Hemoglobin, D292, Gr0: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Hemoglobin, D292, Gr0 | 9 | 5 | 8 | 8 | 15 | 23
  Hemoglobin, D292, Gr1: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  Hemoglobin, D292, Gr1 | 0 | 0 | 0 | 1 | 0 | 0
  Hemoglobin, D315, Gr0: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  Hemoglobin, D315, Gr0 | 16 | 21 | 19 | 18 | 21 | 24
  Hemoglobin, D315, Gr1: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  Hemoglobin, D315, Gr1 | 4 | 0 | 3 | 1 | 0 | 0
  Hemoglobin, D315, Gr2: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  Hemoglobin, D315, Gr2 | 0 | 0 | 0 | 1 | 0 | 0
  Platelets, SCR, Gr0 | 26 | 26 | 26 | 26 | 26 | 24
  Platelets, D36, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Platelets, D36, Gr0 | 26 | 25 | 25 | 26 |  |
  Platelets, D59, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  Platelets, D59, Gr0 | 26 | 25 | 25 | 26 |  |
  Platelets, D204, Gr0: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  Platelets, D204, Gr0 | 23 | 24 | 24 | 25 | 23 |
  Platelets, D227, Gr0: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  Platelets, D227, Gr0 | 23 | 23 | 24 | 24 | 23 |
  Platelets, D292, Gr0: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 22
  Platelets, D292, Gr0 | 9 | 5 | 8 | 8 | 15 | 19
  Platelets, D292, Gr1: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 22
  Platelets, D292, Gr1 | 0 | 0 | 0 | 0 | 0 | 2
  Platelets, D292, Gr2: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 22
  Platelets, D292, Gr2 | 0 | 0 | 0 | 1 | 0 | 0
  Platelets, D292, Gr3: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 22
  Platelets, D292, Gr3 | 0 | 0 | 0 | 0 | 0 | 1
  Platelets, D315, Gr0: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 23
  Platelets, D315, Gr0 | 20 | 21 | 22 | 19 | 21 | 22
  Platelets, D315, Gr1: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 23
  Platelets, D315, Gr1 | 0 | 0 | 0 | 1 | 0 | 1
  WBC Decrease, SCR, Gr0 | 25 | 25 | 26 | 26 | 26 | 24
  WBC Decrease, SCR, Gr1 | 1 | 1 | 0 | 0 | 0 | 0
  WBC Decrease, D36, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  WBC Decrease, D36, Gr0 | 26 | 24 | 25 | 26 |  |
  WBC Decrease, D36, Gr1: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  WBC Decrease, D36, Gr1 | 0 | 1 | 0 | 0 |  |
  WBC Decrease, D59, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  WBC Decrease, D59, Gr0 | 26 | 25 | 24 | 26 |  |
  WBC Decrease, D59, Gr1: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  WBC Decrease, D59, Gr1 | 0 | 0 | 1 | 0 |  |
  WBC Decrease, D204, Gr0: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  WBC Decrease, D204, Gr0 | 23 | 24 | 24 | 25 | 23 |
  WBC Decrease, D227, Gr0: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  WBC Decrease, D227, Gr0 | 23 | 23 | 22 | 24 | 23 |
  WBC Decrease, D227, Gr1: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  WBC Decrease, D227, Gr1 | 0 | 0 | 2 | 0 | 0 |
  WBC Decrease, D292, Gr0: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  WBC Decrease, D292, Gr0 | 8 | 4 | 6 | 8 | 15 | 20
  WBC Decrease, D292, Gr1: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  WBC Decrease, D292, Gr1 | 1 | 1 | 2 | 1 | 0 | 3
  WBC Decrease, D315, Gr0: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  WBC Decrease, D315, Gr0 | 20 | 21 | 21 | 20 | 20 | 24
  WBC Decrease, D315, Gr1: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  WBC Decrease, D315, Gr1 | 0 | 0 | 1 | 0 | 1 | 0
  WBC Increase, SCR, Gr0 | 25 | 26 | 26 | 25 | 25 | 22
  WBC Increase, SCR, Gr1 | 1 | 0 | 0 | 1 | 1 | 2
  WBC Increase, D36, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  WBC Increase, D36, Gr0 | 25 | 25 | 25 | 23 |  |
  WBC Increase, D36, Gr1: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  WBC Increase, D36, Gr1 | 1 | 0 | 0 | 3 |  |
  WBC Increase, D59, Gr0: number analyzed (Participants) | 26 | 25 | 25 | 26 | 0 | 0
  WBC Increase, D59, Gr0 | 26 | 25 | 25 | 26 |  |
  WBC Increase, D204, Gr0: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  WBC Increase, D204, Gr0 | 23 | 24 | 24 | 23 | 21 |
  WBC Increase, D204, Gr1: number analyzed (Participants) | 23 | 24 | 24 | 25 | 23 | 0
  WBC Increase, D204, Gr1 | 0 | 0 | 0 | 2 | 2 |
  WBC Increase, D227, Gr0: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  WBC Increase, D227, Gr0 | 22 | 23 | 23 | 24 | 23 |
  WBC Increase, D227, Gr1: number analyzed (Participants) | 23 | 23 | 24 | 24 | 23 | 0
  WBC Increase, D227, Gr1 | 1 | 0 | 1 | 0 | 0 |
  WBC Increase, D292, Gr0: number analyzed (Participants) | 9 | 5 | 8 | 9 | 15 | 23
  WBC Increase, D292, Gr0 | 9 | 5 | 8 | 9 | 15 | 23
  WBC Increase, D315, Gr0: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  WBC Increase, D315, Gr0 | 19 | 20 | 22 | 20 | 19 | 24
  WBC Increase, D315, Gr1: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  WBC Increase, D315, Gr1 | 0 | 0 | 0 | 0 | 2 | 0
  WBC Increase, D315, Gr2: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  WBC Increase, D315, Gr2 | 0 | 1 | 0 | 0 | 0 | 0
  WBC Increase, D315, Gr3: number analyzed (Participants) | 20 | 21 | 22 | 20 | 21 | 24
  WBC Increase, D315, Gr3 | 1 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Subjects With Any, Fatal or Related SAE, After Challenge
Description: as for outcome 9
Time Frame: From day of challenge (Day 287) to the end of the challenge phase (Day 315)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited adverse events were reported during the 7-day follow-up period and unsolicited adverse events during the 30-day follow-up period after vaccination. Serious adverse events were reported during the whole study period (from Day 1 up to study conclusion at Day 377).
Arm/Group | AduFx Group | 2PedFx Group | PedFx Group | Adu2Fx Group | Adu1Fx Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26 | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26 | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 26/26 | 25/26 | 23/26 | 25/26 | 24/26 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AduFx Group (N=26) | 2PedFx Group (N=26) | PedFx Group (N=26) | Adu2Fx Group (N=26) | Adu1Fx Group (N=26) | Control Group (N=24)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 4 (7) | 3 (4) | 5 (6) | 5 (7) | 0 (0) | 0 (0)
Fatigue (General disorders) | 16 (28) | 20 (33) | 15 (31) | 13 (29) | 14 (20) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 14 (23) | 18 (31) | 12 (19) | 15 (23) | 12 (15) | 0 (0)
Injection site pain (General disorders) | 23 (54) | 23 (49) | 23 (55) | 22 (50) | 20 (34) | 0 (0)
Injection site swelling (General disorders) | 9 (13) | 15 (26) | 9 (14) | 9 (10) | 8 (8) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (10) | 12 (15) | 4 (5) | 5 (6) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 20 (35) | 20 (35) | 18 (28) | 16 (28) | 12 (19) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 9 (12) | 11 (16) | 9 (18) | 6 (7) | 8 (11) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (2) | 2 (4) | 2 (3) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 7 (8) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypobarism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT03162614/Prot_002.pdf
  • Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT03162614/SAP_003.pdf